CLINICAL TRIAL: NCT03883269
Title: A Randomized, Placebo-controlled, Evaluator-blinded, Study to Assess the Anti-inflammatory Effects of Topical Erythromycin and Clindamycin in Patients With Inflammatory Facial Acne
Brief Title: Anti-inflammatory Effects of Topical Erythromycin and Clindamycin in Acne Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Human Drug Research, Netherlands (Other)
Collaborators: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHDR1732
Record Dates: First submitted 2018-02-15; First posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Erythromycin; Clindamycin

STUDY DESIGN:
Intervention Model Description: A randomized, open-label, placebo-controlled, evaluator-blinded study.
Who Masked: Outcomes Assessor
Masking Description: Evaluator-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Erythromycin 4% (Experimental): Erythromycin 4% topical gel formulation, BID, 4 weeks
  Interventions: Drug: Erythromycin 4% topical gel formulation
- Clindamycin 1% (Experimental): Clindamycin 1% topical lotion formulation, BID, 4 weeks
  Interventions: Drug: Clindamycin 1% topical lotion formulation
- ethanol solution (Placebo Comparator): 70% topical ethanol solution, BID, 4 weeks
  Interventions: Drug: 70% topical ethanol solution

INTERVENTIONS:
Drug: Erythromycin 4% topical gel formulation — Erythromycin 4% topical gel formulation, BID, 4 weeks
  Arms: Erythromycin 4%
Drug: Clindamycin 1% topical lotion formulation — Clindamycin 1% topical lotion formulation, BID, 4 weeks
  Arms: Clindamycin 1%
Drug: 70% topical ethanol solution — 70% topical ethanol solution, BID, 4 weeks
  Arms: ethanol solution

SUMMARY:
The combined bacteriostatic and immunomodulatory effects of erythromycin and clindamycin will be explored. Treatment effects will be extensively characterized by conventional methods including lesion counts, global assessment scales and visual grading as well as state-of-the-art methodology, including multi-modal photo analysis, perfusion by laser speckle contrast imaging, analysis of local skin surface, biopsy biomarkers and skin microbiota. This extensive response profiling, combined with the mechanistic insights from concurrent in vitro and in vivo studies in healthy volunteer challenges, will increase the understanding of erythromycin's and clindamycin's effects in acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects, 18 to 45 years of age. The health status is verified by absence of evidence of any clinical significant active or uncontrolled chronic disease other than AV following a detailed medical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, virology and urinalysis;
2. Mild to moderate inflammatory acne vulgaris on the face, ≥5 inflammatory lesions (papules and/or pustules), present at screening and baseline visit
3. A maximum of 5 nodules present at screening and baseline visit
4. Inflammatory acne present for at least 6 months
5. Fitzpatrick skin type I-II (Caucasian)
6. Able and willing to give written informed consent and to comply with the study restrictions.
7. Willing to comply with 2x2mm facial skin punch biopsies

Exclusion Criteria:

1. Severe acne where systemic treatment is needed
2. Use of any topical (anti-acne) medication (prescription or OTC) within 2 weeks prior to baseline
3. Use of any oral/systemic treatment for acne, including oral antibiotics, excluding OAC, within 4 weeks prior to baseline
4. Use of systemic isotretinoin within 6 months prior to baseline
5. History of pathological scar formation (keloid, hypertrophic scar)
6. Known hypersensitivity to erythromycin or clindamycin, drugs of the same class, or any of their excipients.
7. Known contact dermatitis reaction to any product
8. Tanning due to sunbathing, excessive sun exposure or a tanning booth within 3 weeks of enrollment.
9. Participation in an investigational drug or device study within 3 months prior to screening or more than 4 times a year.
10. Loss or donation of blood over 500 mL within three months (males) or four months (females) prior to screening
11. Pregnant, a positive pregnancy test, intending to become pregnant, or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy endpoint 1 - Change in lesion count | Day 0, day 7, day 14, day 21, day 28 and day 42
  The inflammatory lesions include papules pustules and nodules/cysts. At screening and every study visit, the evaluator will count the inflammatory lesions separately by area on the face (forehead, right cheek, left cheek, chin and nose). All lesion counts during the treatment and follow-up period will be performed by a treatment-blinded evaluator
Efficacy endpoint 2 - Change in investigator Global Assessment acne (IGA) | Day 0, day 7, day 14, day 21, day 28 and day 42
  Acne severity will be assessed at screening and every study visit by the Investigator Global Assessment for facial acne (clear, almost clear, mild, moderate, severe, very severe). This will be done by a treatment blinded evaluator.
Change in Patient Reported Outcome (PRO) | Day 0 and day 28
  Pre-dose and at EOT patients will be asked how they would rate their acne that day using the subjective Patient Global Assessment (clear, almost clear, mild, moderate, severe, very severe)
Pharmacodynamic endpoints 1 - Change in Standardized facial photography by Canfield Visia and via selfie app | Day 0, day 7, day 14, day 21, day 28 and day 42
  A standardized set of 3 facial photos (front, left, right) will be taken every study visit by Canfield Visia CR. Furthermore, patients will take daily selfies with a validated mobile app.
Pharmacodynamic endpoints 2 - Change in Sebum measurements by Sebumeter® | Day 0, day 7, day 14, day 21, day 28 and day 42
  Sebum excretion will be measured every study visit by Sebumeter®. The measurement will be repeated for 3 times and the average will be used for the analysis.
Pharmacodynamic endpoints 3 - Change in Perfusion by Laser Speckle Contrast Imaging (LSCI) | Day 0, day 7, day 14, day 21, day 28 and day 42
  Cutaneous microcirculation will be assessed using the laser speckle imager (LSCI; PeriCam PSI System, Perimed Jäfälla, Sweden). Measurements have to be performed in a temperature controlled room with a temperature around 22°C. The subject has to get accommodated to the room temperature for a minimum of 15 minutes prior to testing. After this, the speckle assessments can commence. Briefly, the subject will be resting for at least ten minutes before any measurements take place. A suitable area of the face will be identified. This area will be illuminated' by the laser and the response signal will be captured.
  If no suitable area can be identified, the measurement will not be performed and data will be entered as missing.
Pharmacodynamic endpoints 4 - Change in Morphology by Optical Coherence Tomography (OCT) | Day 0, day 7, day 14, day 21, day 28 and day 42
  Skin morphology will be assessed by optical coherence tomography at every study visit. Optical coherence tomography uses reflected light returning from skin tissue to create an image of the skin and 2 mm below the skin. The visualization can be done because different skin structures reflect light in a different way and can therefore be distinguished. Optical coherence tomography is similar to ultrasound however instead of sound it uses light refraction to visualize tissue.
Pharmacodynamic endpoints 5 - Change in Local skin biopsy biomarkers | Day 0 and day 28
  Two-millimetre punch biopsies are taken at day 0 and day 28 from a papule or pustule. Moreover, at day 0 a biopsy will be taken from nonlesional non-facial skin (upper back) as healthy control. The biopsies will be placed in RNAlater medium directly after harvest of the biopsy and stored at 4°C. Biomarker sequencing will be performed by RNA extraction and quantitative PCR will be performed for a subset of immunomodulatory biomarkers (including but not limited to IL-1b, IL-1a, TNF-a IL-6, IL-12, IL-8, IL-10, IL-17, IFN-g).
Pharmacodynamic endpoints 6 - Change in Local skin surface biomarkers by TAP | Day 0, day 7, day 14, day 21, day 28 and day 42
  Skin biomarkers will be measured pre-dose and after 7, 14, 21, 28, and 42 days by TAP (FibroTx, Estonia). TAP consists of a multiplex capture-antibody micro-array that is supported by a dermal adhesive bandage for fixture to skin. When TAP is applied to skin and left on for 20 minutes, the antibodies printed on the micro-array capture biomarkers from skin through immune recognition.
  Biomarkers (IL-1a, IL-1b, TNF-a, IL-8, IL-6, IL-17) captured from skin by TAP are qualitatively and quantitatively analyzed by spot-ELISA by a specific TAP analyzer.
Pharmacodynamic endpoints 7 - Change in skin microbiota | Day 0, day 7, day 14, day 21, day 28 and day 42
  The skin swab will be placed in a 2 ml lysis tube containing DNA/RNA shield to stabilize and preserve the DNA. The DNA extraction will be performed using adapted DNA extraction method based on the Zymo Research fecal DNA extraction methodology. The microbiome will be analyzed according to 16S rRNA gene sampling
Pharmacodynamic endpoints 8 - Change over time in p. acnes cultures | Day 0, day 7, day 14, day 21, day 28 and day 42
  Swabs of predefined lesional (papule of pustule) and non-lesional skin will be taken with a sterile cotton swab. Colony numbers (colony forming units - CFU) and minimal inhibitory concentrations (MIC) will be reported. In addition, swabs of other lesions (i.e. nodules or scars) may be taken if applicable.
  Moreover, in order to study P. acnes in the pilosebaceous unit a comedo extraction will be performed and the sebum will be cultured for P. acnes. Comedo extraction will be performed if applicable (i.e. if the patient has comedones).
Pharmacodynamic endpoints 9 - Change over time in faecal microbiota | before day 0 and after day 28
  Faecal samples will be collected at home. Subjects will use a 'faeces catcher' in their toilet and afterwards use a cotton swab to transfer a scoop of faeces to a 2 ml lysis tube (REF ZY-R1103, Zymo Research) containing DNA/RNA shield to stabilize and preserve the DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rissmann, PharmD, PhD, Principal Investigator — CHDR
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands